CLINICAL TRIAL: NCT05526846
Title: Introducing a Plant-Based Diet for Patients With Colorectal Diseases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Cindy Kin, Assistant Professor of Surgery, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 66060
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Diet, Healthy; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Invervention group (Experimental): Participants will receive an educational intervention about how to incorporate more plant foods into their diet.
  Interventions: Behavioral: Plant-based diet education

INTERVENTIONS:
Behavioral: Plant-based diet education — Participants will receive weekly emails with information about plant-based diets and a goal/task for each week.
  There will be a 'core curriculum' that will be sent to all participants, as well as additional information according to the participant's stage of change and food choice preferences.
  All information will be available on a website that will be created for this study. The website will feature curated information about plant-based diets, that is tailored to patients who had recent colorectal operations and may have a colostomy or an ileostomy.

SUMMARY:
Dietary patterns are a potentially modifiable risk factor for colon cancer recurrence, flares in inflammatory bowel diseases, and for chronic diseases. Nutritional counseling is rarely brought up during medical appointment. As a result, patients are often left confused regarding which specific dietary recommendation to follow after surgical treatment. A plant-based diet is naturally high in fiber and is beneficial to long-term health, especially for patients with colorectal diseases.

The aims of this study are to:

1. Determine whether an educational intervention is effective in increasing intake of plants
2. Identify barriers and facilitators to adoption of a plant-based diet among patients with colorectal diseases
3. Identify secondary health gains related to adoption of a plant-based diet.

DETAILED DESCRIPTION:
Standard of care: patients with colorectal diseases are sometimes advised to eat healthfully before and after to surgery. They are also encouraged to increase fiber intake and to take fiber supplements, but not particularly encouraged to eat more plants.

Research Activities:

1. Screening: eligible patients will be identified through screening the clinic schedules. Participants that might be eligible will be asked if they are interested in being contacted by the research team.
2. Enrollment: in person or remotely, if the patient demonstrates interest in participating, the research team will explain details about the study. If the patient agrees, they will be asked to provide consent
3. Intervention: at baseline, data will be collected regarding clinical information of the patients (age, body mass index, comorbidities, medications or supplements, physical activity level), and baseline dietary pattern, which will be evaluated through a validated shortened Food Frequency Questionnaire. Patients will be assessed regarding their stage of change according to the transtheoretical model. A Food Choice Questionnaire will be administered to understand what drives their food choices. A Quality of Life questionnaire for patients recovering from surgery will also be administered.

   The intervention proposed is a "6-week challenge", in which participants will be encouraged to make at least one change towards a plant-based diet per week. They will receive weekly emails with information about plant-based diets and a goal/task for each week.

   There will be a 'core curriculum' that will be sent to all participants, as well as additional information according to the participant's stage of change and food choice preferences.

   All information will be available on a website that was created for this study (http://eat2heal.su.domains/). The website features curated information about plant-based diets, and is tailored to patients who had recent colorectal operations and may have a colostomy or an ileostomy. The goal is to recruit 60 patients with colorectal diseases
4. Closeout: At the end of the intervention period, the quality of life and food frequency questionnaires will be re-administered.

Semi-structured interviews will be conducted at the end of the intervention period to identify areas for improvement, barriers and facilitators to adopt a plant-based diet, and other health attitudes that may have changed as a result of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Good English comprehension
* Diagnosis of a colorectal disease
* Must be able to maintain oral nutrition
* Access to Internet and email

Exclusion Criteria:

* Patients who are unable to maintain oral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Effect of the intervention on participant's Healthy Plant-Based Diet Index | 2 weeks after the intervention
  The Healthy Plant-Based Diet Index will be calculated from a standardized Food Frequency Questionnaire, which will be administered upon enrollment and 2 weeks after the end of the intervention

SECONDARY OUTCOMES:
Effect of the intervention on participant's Quality of Life | 2 weeks after the intervention
  Quality of life will be assessed through a validated Quality of Life Questionnaire that will be administered upon enrollment and 2 weeks after the end of the intervention
Barriers and facilitators to transitioning to a healthier diet | 2 weeks after the intervention
  A semi-structured interview will be performed to identify barriers and facilitators to transitioning to a healthier diet
Secondary health gains associated with adopting a plant-based diet | 2 weeks after the intervention
  A semi-structured interview will be performed to identify secondary health gains that may be expected by adopting a plant-based diet

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Health Care, Stanford, California, United States